CLINICAL TRIAL: NCT05044416
Title: Tracheal Intubation With VieScope Versus Videolaryngoscopy in Patients for Elective Surgery With an Expected Difficult Airway - a Prospective Randomized Trial (VieScOP-II)
Brief Title: VieScope in Patients With an Expected Difficult Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VieScOP-II
Record Dates: First submitted 2021-09-05; First posted 2021-09-14 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Airway Management

STUDY DESIGN:
Intervention Model Description: randomized 1:1
Who Masked: Participant
Masking Description: device for intubation may not be blinded for provider or investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VieScope (Experimental): intubation with the VieScope laryngoscope
  Interventions: Device: VieScope
- Videolaryngoscopy (Active Comparator): intubation with videolaryngoscope
  Interventions: Device: Videolaryngoscopy

INTERVENTIONS:
Device: VieScope — intubation with VieScope laryngoscope
  Arms: VieScope
Device: Videolaryngoscopy — intubation with videolaryngoscope
  Arms: Videolaryngoscopy

SUMMARY:
Patients requiring endotracheal intubation for elective surgery with an expected difficult airway are randomized to be intubated either by a) VieScope or b) videolaryngoscopy.

DETAILED DESCRIPTION:
Tracheal intubation is required for different surgical procedures for mechanical ventilation and to prevent aspiration of secretions. In patients with an expected difficult airway, tracheal intubation is often performed by videolaryngoscopy (VL). However, this technique has limitations and may fail due to insufficient visualization of the larynx. A new device has been introduced that consists of an illuminated straight plastic tube for laryngoscopy (VSC, Vie Scope, Adroit Surgical, Oklahoma City, OK, USA) that enables for indirect intubation over a stylet.

So far, the VSC has shown promising results in manikin studies for intubation in normal and difficult airways. We aim to test the VSC in patients compared to videolaryngoscopy in a prospective randomized non-inferiority trial.

Patients will be assessed for eligibility in the Anesthesiology Pre-assessment Clinic of the University Medical Center Hamburg-Eppendorf prior to elective surgery. All patients receive a structured preoperative airway assessment.

Patients are randomized 1:1 to either intervention or control group. Patients randomized to the intervention group will be intubated with the VSC. Patients randomized to the control group are intubated with a MacIntosh type videolaryngoscope (CMAC, Storz, Germany).

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring general anesthesia with transoral tracheal intubation for elective surgery
* Age ≥ 18
* Preoperative airway assessment reveals an expected difficult airway (rated by the responsible anesthetist in the Pre-assessment Clinic based on the existing in-house algorithm)

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Confirmed indications for awake fiberoptic intubation especially due to enoral, pharyngeal tumors, abscesses or other processes
* Planned endotracheal intubation without deep anesthesia or neuromuscular blocking agents (e.g. awake videolaryngoscopy)
* Required transnasal tracheal intubation (e.g. for surgical reasons)
* Requirement of special endotracheal tubes such as laser or RAE tubes for surgical reasons
* Patients at risk for pulmonary aspiration who qualify for rapid sequence induction
* Loose teeth
* Denial of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-09-11 (Actual); Primary Completion 2022-06-26 (Actual); Study Completion 2022-06-26 (Actual)

PRIMARY OUTCOMES:
Percentage of Glottis Opening (POGO) scale | 15 min
  intubating conditions according to the percentage of glottis opening scale (POGO), range 0-100%, higher values better

SECONDARY OUTCOMES:
first attempt success rate | 15 min
  percentage of successful intubations with one attempt
time to intubation | 15 min
  time until tracheal airway access is established
Cormack-Lehane | 15 min
  intubating conditions according to Cormack-Lehane
overall success rate | 15 min
  percentage of successful intubations with the allocated procedure
time to successful intubation with one attempt | 15 min
  time until tracheal airway access is established in patients that are intubated at first attempt
intubation difficulty | 15 min
  subjective rating on a visual analogue scale (0-100, higher values indicate more difficult intubation) of the difficulty of airway management and questionnaire
number of attempts | 15 min
  total number of attempts until airway established
aspiration | 15 min
  percentage of patients that vomit and aspirate during intubation
esophageal intubation | 15 min
  percentage of accidental esophageal intubation attempts
hypoxia | 15 min
  percentage of patients with a desaturation below a pulsoximetric saturation of 80%
hypotension | 15 min
  percentage of patients with a systolic blood pressure below 70 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Joern Grensemann, MD, Study Chair — Universitätsklinikum Hamburg-Eppendorf; Martin Petzoldt, MD, Study Chair — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Petzoldt M, Grun C, Wunsch VA, Bauer M, Hardel TT, Grensemann J. Vie Scope(R) versus videolaryngoscopy in expected difficult airways: a randomized controlled trial. Can J Anaesth. 2023 Sep;70(9):1486-1494. doi: 10.1007/s12630-023-02534-y. Epub 2023 Aug 3. PMID 37537324